CLINICAL TRIAL: NCT04851184
Title: Dose of Vestibular Rehabilitation Required for Clinical Improvements in Individuals With Vestibular Hypofunction.
Brief Title: Dose of Vestibular Rehabilitation for Vestibular Hypofunction
Acronym: VRVR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment challenges for in-person visits of the affected population and a change in employment of the study team
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Keith Cole, Assistant Professor, George Washington University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCR180548
Record Dates: First submitted 2021-04-11; First posted 2021-04-20 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Vestibular Disorder
Keywords: gaze stability; vestibular hypofunction
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Usual Vestibular Rehabilitation Care (Active Comparator): Participants in this arm will perform typical PT in the clinic and home environment. They will be asked to keep a log to track their HEP.
  Interventions: Behavioral: Gaze stabilization non-instrumented
- Home Exercises Using Virtual Reality Device (Experimental): Participants in this arm will perform typical PT in the clinic, but will use the virtual reality device as part of their HEP.
  Interventions: Device: Gaze stabilization Exercises using Virtual Reality Device
- Healthy Control (No Intervention): Age-matched healthy control subjects will perform all balance, gait, vestibular, and patient reported outcome measure assessments, including performing 30 seconds of each level of gaze stability exercise for an active comparison to outcomes obtained to those with vestibular disorders. The healthy-control group will only be assessed at baseline (a single visit).

INTERVENTIONS:
Device: Gaze stabilization Exercises using Virtual Reality Device — Participants will utilize a wireless virtual reality headset to perform their gaze stabilization exercises to better control the background and visual field as well as collect data related to speed, excursion, and duration of head movements.
  Arms: Home Exercises Using Virtual Reality Device
Behavioral: Gaze stabilization non-instrumented — Participants will perform gaze stabilization exercises in a non-instrumented manner. Subjects are instructed to focus on a letter on a piece of paper held at arm's length. They are instructed to move their head back and forth as quickly as they can while keeping the letter in focus. The total duration of the exercise (from 10 - 240 seconds) and background complexity (simple to complex moving) are increased gradually according to patient symptoms.
  Arms: Usual Vestibular Rehabilitation Care

SUMMARY:
The purposes of this research are to 1) utilize virtual reality (VR) to evaluate the exercise dose required to improve symptoms in those with vestibular (dizziness) disorders, 2) compare VR vestibular exercises to standard exercises, and 3) compare exercise performance outcomes to healthy controls without vestibular disorders. Even though more than 35% of those over 40, and ~50% of those who have had concussion have such symptoms, the dose of specific exercises targeted to improve symptoms is not well defined. In this study, the investigators will use a wireless VR device to measure key parameters and response to exercise. Another advantage of the VR device is the ability to control what the individual can see while performing the exercise. In normal daily life, moving objects and distracting backgrounds can make vestibular exercise too uncomfortable to perform. Using these methods, the investigators aim to determine the appropriate type and amount of exercise required for symptom improvement. This study will also compare the effectiveness of performing exercises in the virtual reality environment to standard physical therapy and to healthy persons without history of vestibular disorders. Three categories of vestibular disorders will be investigated with an instrumented and usual therapy group of 1) Unilateral hypofunction, 2) bilateral hypofunction, and 3) post-concussion.

DETAILED DESCRIPTION:
Disorders of vestibular function are prevalent disorders that result in dizziness, decreased balance, and a 12-fold increased risk of falls.1 It has been determined that 20% of community-dwelling adults over the age of 60 report vestibular symptoms prompting a medical evaluation or intervention over a one year period.2 This equates to approximately $50.0 billion in annual healthcare costs.3 In the US alone, there are approximately 1.6-3.8 million sport concussions each year,4,5 where 50% of concussed athletes have at least one vestibular type symptom.6 Although the impact of cost has been demonstrated in older adults, the costs of concussion-related dizziness is much more difficult to calculate due simultaneously treating symptoms from multiple systems.

A common treatment for symptoms related to disorders of vestibular function is vestibular rehabilitation, a sub-specialty of physical therapy. These exercises are performed daily by Subjects at home and consist of visually fixating on a target while moving the head and/or the object on which the subject is fixating. To alter exercise difficulty, exercise parameters are altered including: visual background complexity (plain and dark, busy but stationary, moving objects, rapidly moving objects), postural positioning (seated, standing with a wide base of support, standing with a narrow base of support, standing on one leg), and duration of exercise (from 5 seconds to approximately 2 minutes). Early evidence shows that vestibular rehabilitation exercises provided by a physical therapist is an effective method of ameliorating vestibular hypofunction. Further, effectiveness of vestibular rehabilitation does not decline with increasing age of the patient,8 indicating benefit for all ages that are affected. Unfortunately, many factors limit the ability to determine efficiency and efficacy of treatment and have been highlighted in a recent clinical practice guideline9 and systematic review5,10. Limitations include: poor measurement of prescribed exercise compliance by depending on subjective report, inability to control for environmental factors during home program execution, and the influence of noxious vestibular input associated with traveling to attend scheduled physical therapy visits. These factors hinder performing high quality efficacy studies, resulting in exercise prescription being largely based on expert opinion, the lowest level on the hierarchy of evidence-based practice.11 In fact, current opinion indicates that exercises should be performed 3 times a day for a total of 12 minutes with each bout lasting approximately 2 minutes, all with no clear indication of speed and amplitude of performance. In this study, the investigators aim to use a commercially available virtual reality device to deliver usual vestibular rehabilitation exercises, while using the device's inbuilt sensors to accurately measure head movement, speed and duration. Using this device, the investigators will assess compliance and dose of exercises required to reduce symptoms of dizziness and imbalance and to determine if performing such exercises in a virtual reality environment will provide similar results to that usual rehabilitation techniques.

When a potential subject is identified, the subject will be screened for appropriateness of inclusion for this study. After informed consent has been obtained from a recruited subject, those with Unilateral Vestibular Hypofunction (UVH) will be asked to perform a 4-week intervention, while those with Bilateral Vestibular Hypofunction (BVH) or those post-concussion will each be asked to perform a 12-week intervention. Those with UVH will undergo a shorter intervention due to strong evidence that neural adaptation occurs much more quickly (usually 4 weeks) than those with BVH and history of concussion.9,10,17-19 The intervention will consist of physical therapy visits combined with a home program of specific vestibular exercises. Each subject will be asked to attend physical therapy visits at least one time per week throughout the 4- or 12-week period.

Assessments will be performed on all groups and consist of a combination of vestibulo-ocular assessment, balance and clinical functional outcome measures, and surveys of subject satisfaction. Subjects are randomly assigned to the usual rehabilitation or intervention group based on each of the following diagnostic categories.

The compliance to exercises will be obtained from a log in the virtual reality device for the VR group, and will be paper based for the usual physical therapy group. Subjects in the three intervention groups will be asked to perform the same type of exercises as the usual rehabilitation group, but using a virtual reality device that will be issued to the patient for home use. Subjects will use a custom designed program to perform the exercises using a commercially available virtual reality device (no specialized hardware or additions to the commercially available device will be performed). Subjects will be instructed on the first day in how to operate the Virtual Reality Vestibular Rehabilitation (VRVR) program and how to properly perform the exercises. The VRVR device and software will simulate a virtual reality 'room' with an 'X' fixed in front of a wall. There are six different background complexities. Exercise sessions will start seated upright in a chair and will progress to standing per the home exercise protocol. The system will prompt the patient to begin the exercise and will automatically log the frequency and duration of exercise performed. The system will ask the patient to rate the severity of their symptoms on a 0-10 scale before and after each bout of exercise. Subjects' instruction regarding initial dose and progression will be identical to those given in the usual rehabilitation group. Subjects will be asked to bring their device with them to their 4 week, 8 week, and 12 weeks appointment to transfer their de-identified data and to insure integrity of the data and device. Subjects will be asked to return the device at the end of the intervention period.

Per patient and therapist discretion, additional physical therapy visits may be scheduled to aid in patient understanding of exercise progression protocol, assess correct performance of exercise (with or without virtual reality device). Non-study related physical therapy visits may be scheduled between sessions in order to address impairments unrelated to vestibulo-ocular deficits. These may include interventions to address musculoskeletal deficits or other balance related impairments. Any additional sessions of physical therapy will be reported in order to determine possible confounding information.

There will be an additional group of healthy control subjects that will be tested for only one day. Healthy subjects will be recruited through flyers, approved email lists, and word of mouth in the general public. This healthy control group will perform the same tests as the other groups perform on Day 1. This group will be used to compare outcomes of usual rehabilitation and intervention groups, to the function of those without disorders of vestibular function.

ELIGIBILITY:
Inclusion Criteria:

* Known or suspected vestibular dysfunction
* Healthy volunteers without dizziness to serve as healthy control subjects

Exclusion Criteria:

* Previous cerebrovacular accident (stroke)
* Reported neurologic or oculuomotor disease
* Taking of medications that affect the vestibular or oculomotor system.
* Current symptoms of benign paroxysmal positional hypofunction
* Concussion occuring less than 7 days prior to enrollment in this study
* Currently pregnant, or plan to become pregnant during the timeline of the study
* Chronic kidney disease
* COPD
* Known coronary artery disease or cardiomyopathy
* immunocompromised state from a solid organ transplant
* Severe Obesity as defined by BMI of greater than or equal to 40 kg/m2
* Sickle cell disease

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Goodman, DPT, Principal Investigator — The George Washington University
Locations (1):
- The George Washington University, Department of Health, Human Function and Rehabilitation Science, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agrawal Y, Carey JP, Della Santina CC, Schubert MC, Minor LB. Disorders of balance and vestibular function in US adults: data from the National Health and Nutrition Examination Survey, 2001-2004. Arch Intern Med. 2009 May 25;169(10):938-44. doi: 10.1001/archinternmed.2009.66. PMID 19468085
- [Background] Sloane PD, Coeytaux RR, Beck RS, Dallara J. Dizziness: state of the science. Ann Intern Med. 2001 May 1;134(9 Pt 2):823-32. doi: 10.7326/0003-4819-134-9_part_2-200105011-00005. PMID 11346317
- [Background] Florence CS, Bergen G, Atherly A, Burns E, Stevens J, Drake C. Medical Costs of Fatal and Nonfatal Falls in Older Adults. J Am Geriatr Soc. 2018 Apr;66(4):693-698. doi: 10.1111/jgs.15304. Epub 2018 Mar 7. PMID 29512120
- [Background] Murray DA, Meldrum D, Lennon O. Can vestibular rehabilitation exercises help patients with concussion? A systematic review of efficacy, prescription and progression patterns. Br J Sports Med. 2017 Mar;51(5):442-451. doi: 10.1136/bjsports-2016-096081. Epub 2016 Sep 21. PMID 27655831
- [Background] Kontos AP, Elbin RJ, Schatz P, Covassin T, Henry L, Pardini J, Collins MW. A revised factor structure for the post-concussion symptom scale: baseline and postconcussion factors. Am J Sports Med. 2012 Oct;40(10):2375-84. doi: 10.1177/0363546512455400. Epub 2012 Aug 16. PMID 22904209
- [Background] Alghadir AH, Iqbal ZA, Whitney SL. An update on vestibular physical therapy. J Chin Med Assoc. 2013 Jan;76(1):1-8. doi: 10.1016/j.jcma.2012.09.003. Epub 2012 Dec 26. PMID 23331774
- [Background] Whitney SL, Wrisley DM, Marchetti GF, Furman JM. The effect of age on vestibular rehabilitation outcomes. Laryngoscope. 2002 Oct;112(10):1785-90. doi: 10.1097/00005537-200210000-00015. PMID 12368616
- [Background] Hall CD, Herdman SJ, Whitney SL, Cass SP, Clendaniel RA, Fife TD, Furman JM, Getchius TS, Goebel JA, Shepard NT, Woodhouse SN. Vestibular Rehabilitation for Peripheral Vestibular Hypofunction: An Evidence-Based Clinical Practice Guideline: FROM THE AMERICAN PHYSICAL THERAPY ASSOCIATION NEUROLOGY SECTION. J Neurol Phys Ther. 2016 Apr;40(2):124-55. doi: 10.1097/NPT.0000000000000120. PMID 26913496
- [Background] McDonnell MN, Hillier SL. Vestibular rehabilitation for unilateral peripheral vestibular dysfunction. Cochrane Database Syst Rev. 2015 Jan 13;1(1):CD005397. doi: 10.1002/14651858.CD005397.pub4. PMID 25581507
- [Background] Mantzoukas S. A review of evidence-based practice, nursing research and reflection: levelling the hierarchy. J Clin Nurs. 2008 Jan;17(2):214-23. doi: 10.1111/j.1365-2702.2006.01912.x. Epub 2007 Apr 5. PMID 17419779
- [Background] Cohen HS, Kimball KT. Increased independence and decreased vertigo after vestibular rehabilitation. Otolaryngol Head Neck Surg. 2003 Jan;128(1):60-70. doi: 10.1067/mhn.2003.23. PMID 12574761
- [Background] Bergeron M, Lortie CL, Guitton MJ. Use of Virtual Reality Tools for Vestibular Disorders Rehabilitation: A Comprehensive Analysis. Adv Med. 2015;2015:916735. doi: 10.1155/2015/916735. Epub 2015 Apr 30. PMID 26556560
- [Background] Micarelli A, Viziano A, Augimeri I, Micarelli D, Alessandrini M. Three-dimensional head-mounted gaming task procedure maximizes effects of vestibular rehabilitation in unilateral vestibular hypofunction: a randomized controlled pilot trial. Int J Rehabil Res. 2017 Dec;40(4):325-332. doi: 10.1097/MRR.0000000000000244. PMID 28723718
- [Background] Rosiak O, Krajewski K, Woszczak M, Jozefowicz-Korczynska M. Evaluation of the effectiveness of a Virtual Reality-based exercise program for Unilateral Peripheral Vestibular Deficit. J Vestib Res. 2018;28(5-6):409-415. doi: 10.3233/VES-180647. PMID 30714985
- [Background] Alahmari KA, Sparto PJ, Marchetti GF, Redfern MS, Furman JM, Whitney SL. Comparison of virtual reality based therapy with customized vestibular physical therapy for the treatment of vestibular disorders. IEEE Trans Neural Syst Rehabil Eng. 2014 Mar;22(2):389-99. doi: 10.1109/TNSRE.2013.2294904. PMID 24608691
- [Background] Hillier SL, McDonnell M. Vestibular rehabilitation for unilateral peripheral vestibular dysfunction. Clin Otolaryngol. 2011 Jun;36(3):248-9. doi: 10.1111/j.1749-4486.2011.02309.x. No abstract available. PMID 21752206
- [Background] Cohen HS, Gottshall KR, Graziano M, Malmstrom EM, Sharpe MH, Whitney SL; Barany Society Ad Hoc Committee on Vestibular Rehabilitation Therapy. International guidelines for education in vestibular rehabilitation therapy. J Vestib Res. 2011;21(5):243-50. doi: 10.3233/VES-2011-0424. PMID 22101295

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 31 healthy controls were approached, and 28 healthy controls were enrolled in and completed the study. Three potential participants were excluded due to not meet the entry criterion of sufficient convergence (as determined by the oculomotor screening). No subjects were approached or recruited into the usual vestibular rehabilitation care, nor the home exercises using virtual reality device arms, due to the departure of study personnel able to recruit the stated populations.
Groups:
- Healthy Control: Age-matched healthy control subjects will perform all balance, gait, vestibular, and patient reported outcome measure assessments, including performing 30 seconds of each level of gaze stability exercise for an active comparison to outcomes obtained to those with vestibular disorders. Healthy control participants will only be assessed at baseline (a single visit).
Period: Overall Study
Arm/Group | Healthy Control | Usual Vestibular Rehabilitation Care | Home Exercises Using Virtual Reality Device
Started | 28 | 0 | 0
Completed | 28 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Recruitment issues resulted in zero participants in two arms of the study before the study was terminated early.
Groups:
- Healthy Control: Age-matched healthy control subjects will perform all balance, gait, vestibular, and patient reported outcome measure assessments, including performing 30 seconds of each level of gaze stability exercise for an active comparison to outcomes obtained to those with vestibular disorders.
- Total: Total of all reporting groups
Arm/Group | Healthy Control | Usual Vestibular Rehabilitation Care | Home Exercises Using Virtual Reality Device | Total
Number analyzed (Participants) | 28 | 0 | 0 | 28
Age, Continuous [Mean (Full Range); unit: Years] | 23 [22 to 61] |  |  | 23 [22 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 0 | 0 | 20
  Male | 8 | 0 | 0 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Dizziness Handicap Inventory [Median (Full Range); unit: unit on a scale] — The Dizziness Handicap Inventory (DHI) is a 25-item questionnaire used to measure a patient's self-perceived impact of dizziness on their daily life, divided into physical, emotional, and functional subscales. In this study, only the total score (sum of subscales) was used. To score the DHI, each of the 25 questions is answered with "Yes" (4 points), "Sometimes" (2 points), or "No" (0 points), resulting in a total score from 0 to 100. A higher score indicates a greater perceived handicap, a lower score indicates less perceived handicap.
  unit on a scale | 29 [28 to 30] |  |  | 29 [28 to 30]
Head Impulse Test [Count of Participants; unit: Participants] — The head impulse test (HIT) assesses the vestibulo-ocular reflex (VOR) to detect peripheral vestibular dysfunction, or a weakened balance system in the inner ear. In the test, the examiner quickly rotates a patient's head while the patient tries to keep their eyes fixed on a target. A normal response involves the eyes staying fixed on the target, but an abnormal test shows the eyes moving away with the head and then quickly "catching up" with a corrective saccade, indicating the VOR isn't keeping up. Count of participants enrolled in the study are those with a positive clinical finding.
  Participants | 0 |  |  | 0
Visual Vertigo Analogue Scale [Mean (Full Range); unit: units on a scale] — The Visual Vertigo Analogue Scale (VVAS) is a 9-item self-administered questionnaire that assesses the intensity of visual vertigo in various challenging visual situations. Patients mark a 10-cm line for each of the nine items to indicate dizziness severity (0 indicates no dizziness and 10 as extreme). Scores are averaged and then multiplied by 10 for a scale from 0 to 100, where a lower score indicates a milder symptom level, and higher score indicates more severe symptoms of visual vertigo.
  units on a scale | 0.23 [0 to 3] |  |  | 0.23 [0 to 3]
Functional Gait Assessment [Median (Full Range); unit: Units on a scale] — The Functional Gait Assessment (FGA) is a 10-item clinical test used to assess postural stability during walking and assesses an individual's ability to perform multiple motor tasks while walking. Each of the 10 items is scored on a 0-3 scale (0=severe impairment, 3=normal), with the total score ranging from 0 to 30 indicating balance and gait ability. A higher FGA score signifies better performance, and a lower score indicates poorer performance.
  Units on a scale | 29 [28 to 30] |  |  | 29 [28 to 30]
Modified Clinical Test of Sensory Integration and Balance (mCTSIB) [Median (Full Range); unit: units on a scale] — The Modified Clinical Test of Sensory Integration and Balance (mCTSIB) is a four-condition balance assessment that evaluates how well individuals use their visual, somatosensory, and vestibular systems to maintain balance. The scoring involves timing up to three trials of each of the four conditions for 30 seconds, and then summing the average of trials within each condition. The total score ranges from 0 to 120, where a lower score indicates poorer performance and a higher score indicates better performance.
  units on a scale | 120 [120 to 120] |  |  | 120 [120 to 120]

OUTCOME MEASURES:

1. Primary Outcome: Dizziness Handicap Inventory
Description: Final score on the Dizziness Handicap Inventory. The Dizziness Handicap Inventory (DHI) is a 25-item questionnaire used to measure a patient's self-perceived impact of dizziness on their daily life, divided into physical, emotional, and functional subscales. In this study, only the total score (sum of subscales) was used. To score the DHI, each of the 25 questions is answered with "Yes" (4 points), "Sometimes" (2 points), or "No" (0 points), resulting in a total score from 0 to 100. A higher score indicates a greater perceived handicap, a lower score indicates less perceived handicap. This measure is assessed from 0 to 12 weeks in Intervention Arms; Assessed at a single Baseline timepoint for Healthy Controls.
Time Frame: This measure is assessed from 0 to 12 weeks in Intervention Arms; Assessed at a single Baseline timepoint for Healthy Controls.
Population: Only healthy controls were enrolled in this study due to early termination.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Usual Vestibular Rehabilitation Care | Home Exercises Using Virtual Reality Device | Healthy Control
Number analyzed (Participants) | 0 | 0 | 28
units on a scale |  |  | 29 [28 to 30]

2. Primary Outcome: Head Impulse Test at Final Assessment
Description: Assessment of VOR-evoked gaze stability. The head impulse test (HIT) assesses the vestibulo-ocular reflex (VOR) to detect peripheral vestibular dysfunction, or a weakened balance system in the inner ear. In the test, the examiner quickly rotates a patient's head while the patient tries to keep their eyes fixed on a target. A normal response involves the eyes staying fixed on the target, but an abnormal test shows the eyes moving away with the head and then quickly "catching up" with a corrective saccade, indicating the VOR isn't keeping up. Count of participants enrolled in the study are those with a positive clinical finding. This measure is assessed from 0 to 12 weeks in Intervention Arms; Assessed at a single Baseline timepoint for Healthy Controls.
Time Frame: as for outcome 1
Population: No positive findings in head impulse test was determined due to healthy control individuals only attending one session. Only healthy controls were enrolled in this study due to early study termination.
Measure: Number; unit: Participants with positive findings.
Arm/Group | Usual Vestibular Rehabilitation Care | Home Exercises Using Virtual Reality Device | Healthy Control
Number analyzed (Participants) | 0 | 0 | 28
Participants with positive findings. |  |  | 0

3. Secondary Outcome: Visual Vertigo Analogue Scale Final Assessment
Description: Final assessment. The Visual Vertigo Analogue Scale (VVAS) is a 9-item self-administered questionnaire that assesses the intensity of visual vertigo in various challenging visual situations. Patients mark a 10-cm line for each of the nine items to indicate dizziness severity (0 indicates no dizziness and 10 as extreme). Scores are averaged and then multiplied by 10 for a scale from 0 to 100, where a lower score indicates a milder symptom level, and higher score indicates more severe symptoms of visual vertigo. This measure is assessed from 0 to 12 weeks in Intervention Arms; Assessed at a single Baseline timepoint for Healthy Controls.
Time Frame: as for outcome 1
Population: Only healthy control participants were enrolled due to early termination of this study.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Healthy Control | Usual Vestibular Rehabilitation Care | Home Exercises Using Virtual Reality Device
Number analyzed (Participants) | 28 | 0 | 0
units on a scale | 0.23 [0 to 3] |  |

4. Secondary Outcome: Functional Gait Assessment Final Assessment
Description: The Functional Gait Assessment (FGA) is a 10-item clinical test used to assess postural stability during walking and assesses an individual's ability to perform multiple motor tasks while walking. Each of the 10 items is scored on a 0-3 scale (0=severe impairment, 3=normal), with the total score ranging from 0 to 30 indicating balance and gait ability. A higher FGA score signifies better performance, and a lower score indicates poorer performance. This measure is assessed from 0 to 12 weeks in Intervention Arms; Assessed at a single Baseline timepoint for Healthy Controls.
Time Frame: as for outcome 1
Population: Only healthy control participants were enrolled in this study due to early termination.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Healthy Control | Usual Vestibular Rehabilitation Care | Home Exercises Using Virtual Reality Device
Number analyzed (Participants) | 28 | 0 | 0
units on a scale | 29 [28 to 30] |  |

5. Secondary Outcome: Modified Clinical Test of Sensory Integration and Balance (mCTSIB) Final Performance
Description: The Modified Clinical Test of Sensory Integration and Balance (mCTSIB) is a four-condition balance assessment that evaluates how well individuals use their visual, somatosensory, and vestibular systems to maintain balance. The scoring involves timing up to three trials of each of the four conditions for 30 seconds, and then summing the average of trials within each condition. The total score ranges from 0 to 120, where a lower score indicates poorer performance and a higher score indicates better performance. This measure is assessed from 0 to 12 weeks in Intervention Arms; Assessed at a single Baseline timepoint for Healthy Controls.
Time Frame: as for outcome 1
Population: Only healthy control participants were recruited due to early study termination.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Healthy Control | Usual Vestibular Rehabilitation Care | Home Exercises Using Virtual Reality Device
Number analyzed (Participants) | 28 | 0 | 0
units on a scale | 120 [120 to 120] |  |

ADVERSE EVENTS:
Time Frame: A single visit for healthy controls and for those with vestibular dysfunction from enrollment to the end of the 12-week follow-up.
Description: Those at risk for adverse events in the two intervention arms are due to a lack of participant recruitment before early study termination.
Arm/Group | Healthy Control | Usual Vestibular Rehabilitation Care | Home Exercises Using Virtual Reality Device
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/28 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The intervention's effect cannot be determined because the study terminated early before recruiting adequate intervention groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-13): https://cdn.clinicaltrials.gov/large-docs/84/NCT04851184/Prot_SAP_000.pdf